CLINICAL TRIAL: NCT01845285
Title: A Registry to Evaluate the Direct Flow Medical Transcatheter Aortic Valve System for the Treatment of Patients With Severe Aortic Stenosis
Brief Title: A Registry to Evaluate the Direct Flow Medical Transcatheter Aortic Valve System
Acronym: DISCOVER
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Direct Flow Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: RP 001
Record Dates: First submitted 2013-04-30; First posted 2013-05-03 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Aortic Valve Stenosis
Keywords: transcatheter valve replacement; aortic valve disease; aortic stenosis; Aortic regurgitation,catheter; Effective orifice area
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Valve Disease; Aortic Valve Insufficiency | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- aortic valve disease: aortic valve replacement
  Interventions: Device: Aortic Valve Replacement

INTERVENTIONS:
Device: Aortic Valve Replacement — Transthoracic Echo (TTE),CT Scan (ECG triggered, contrast enhanced),Aorto-Iliac Angiogram,Peripheral Evaluation,Coronary Evaluation,12 lead ECG,Arrhythmia Assessment, New York Heart Association (NYHA) functional status, Modified Rankin Score Assessment (mRS) if symptomatic for stroke, Current Cardiac Medications, Transthoracic echo (TTE)
  Other Names: Direct Flow Medical Percutaneous Aortic Valve 18F System; Discover; Transcatheter

SUMMARY:
The purpose of this postmarket Registry is to assess the standard of care and clinical outcomes of the Direct Flow Medical Transcatheter Aortic Valve System used in clinical routine according to the approved commercial indications. Procedures and assessments required by this registry are generally considered standard of care for Transcatheter Aortic Valve Replacement patients.

Evaluation criteria will be the incidence of mortality/morbidity and adverse events clinical performance, and hemodynamic performance of the DEVICE via ultrasound (echo) and angiographic imaging.

DETAILED DESCRIPTION:
The patient population will include patients who are candidates for transcatheter aortic valve replacement (TAVR). According to routine practice, the heart team (interventional cardiologist and cardiothoracic surgeon) makes a choice to use the Direct Flow Medical Aortic Valve System, compared to other available TAVR prostheses, on the basis of clinical and surgical considerations. Therefore, the valve is implanted when the heart team decides that this product is best suited to the specific patient.

In order to be enrolled in this Registry, the patient must be a candidate for the implantation of the Direct Flow Medical Transcatheter Aortic Valve System, based on the commercial indications as stated in the Instructions for Use.

Therefore, candidates for this study must meet the following criteria (Indications for Use):

1. Age > 70 years old
2. Severe aortic valve stenosis determined by echocardiogram and Doppler:

   * mean gradient >40 mmHg or peak jet velocity >4.0 m/s AND
   * aortic valve area ≤0.8 cm2 or aortic valve area index ≤0.5 cm2/m2
3. Symptomatic aortic valve stenosis (angina, congestive heart failure, NYHA Functional Class ≥ II, or syncope).
4. Patient is an extreme risk candidate for open surgical aortic valve repair such that the site Investigators (interventional cardiologist and cardiothoracic surgeon) agree that medical factors preclude operation, based on the conclusion that the probability of death or serious morbidity exceeds the probability of meaningful improvement due to the patient's co-morbidities (such as, but not limited to, severe COPD, porcelain aorta, previous thorax irradiation) or logistic EuroSCORE ≥ 20.

All the Registry clinical evaluations and tests performed are generally considered standard of care for TAVR patients. When these recommendations conflict with the standard of care at the Registry site, the standard of care should prevail. In addition to the standard of care, the Sponsor recommends one brief additional evaluation (the EQ-5D quality of life measure) be conducted. Failure to perform this evaluation shall not be considered a protocol deviation.

Baseline Clinical Evaluation

* Medical History and Physical Exam
* 12 lead ECG and Arrhythmia Assessment
* Logistic EuroSCORE/STS Score
* New York Heart Association (NYHA) functional status
* Modified Rankin Score Assessment (mRS)
* Current Cardiac Medications Baseline Imaging Studies
* Transthoracic Echo (TTE)
* CT Scan (ECG triggered, contrast enhanced)
* Aorto-Iliac Angiogram:

  1. Peripheral Evaluation
  2. Coronary Evaluation

All patients will have clinical follow-up at hospital discharge, 30 days, 12 months and annually to 3 years and undergo the following evaluations:

* Physical Exam
* 12 lead ECG and Arrhythmia Assessment
* New York Heart Association (NYHA) functional status
* Modified Rankin Score Assessment (mRS) if symptomatic for stroke
* Current Cardiac Medications
* Transthoracic echo (TTE) Patients in whom the heart team has planned to use the Direct Flow Medical Transcatheter Aortic Valve System valve, are informed of the DISCOVER Registry and their consent to participate is required. This study intends to monitor the clinical condition of the patient for a period of 3 years after the operation. By agreeing to participate, the patient agrees to undergo clinical assessments and specific tests at certain intervals (prior to the procedure; during the implantation; at hospital discharge, at 30 days after the procedure, and at 1 year, 2 and 3 years later); the patient also agrees to the collection of these daThe purpose of this Registry is to monitor outcomes data for the Direct Flow Medical Transcatheter Aortic Valve System in the Post Market phase. The primary outcome of interest is freedom from all-cause mortality at 30 days. The results from the pivotal CE mark study (IP 010) yielded a 30 day freedom from all-cause mortality rate of 97%. Should the "true" rate be 97%, then N=250 patients would provide an estimate of the rate with a margin of error of 2%, with 95% confidence.

ELIGIBILITY:
Candidates for this study must meet all of the Indications criteria and none of the Contraindications.

Inclusion Criteria (Indications):

1. Age > 70 years old
2. Severe aortic valve stenosis determined by echocardiogram and Doppler:

   * mean gradient >40 mmHg or peak jet velocity >4.0 m/s
   * aortic valve area ≤0.8 cm2 or aortic valve area index ≤0.5 cm2/m2
3. Symptomatic aortic valve stenosis (angina, congestive heart failure, NYHA Functional Class ≥ II, or syncope).
4. Patient is an extreme risk candidate for open surgical aortic valve repair such that the site Investigators (interventional cardiologist and cardiothoracic surgeon) agree that medical factors preclude operation, based on the conclusion that the probability of death or serious morbidity exceeds the probability of meaningful improvement due to the patient's co-morbidities (such as, but not limited to, severe COPD, porcelain aorta, previous thorax irradiation) or logistic EuroSCORE ≥ 20.

Exclusion Criteria (Contraindications):

The Direct Flow Medical device is contraindicated for post implant balloon valvuloplasty.

Min Age: 71 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The Direct Flow Medical Transcatheter Aortic Valve System is intended for use in patients with severe aortic valve stenosis who require replacement of their native aortic valve but are extreme risk candidates for open surgical replacement. This is in accordance with the product Intended Use in the commercial Instructions for Use.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2013-03; Primary Completion 2016-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Freedom from all-cause mortality at 30 days | 30 days

SECONDARY OUTCOMES:
Device Success (VARC defined) | 30 days
  * Absence of procedural mortality AND
  * Correct positioning of a single prosthetic heart valve into the proper anatomic location AND
  * Intended performance of the prosthetic heart valve (no prosthesis-patient mismatch and mean aortic valve gradient <20mmHg or peak velocity <3m/s, AND no moderate or severe prosthetic valve regurgitation)
Early Safety | 30 days
  * All-cause mortality
  * All stroke (disabling and non-disabling)
  * Life-threatening bleeding
  * Acute Kidney Injury - Stage 2 or 3 (including renal replacement therapy)
  * Coronary artery obstruction requiring intervention
  * Major vascular complications
  * Valve-related dysfunction requiring repeat procedure (BAV, TAVR, or SAVR)
Clinical efficacy | 30 days through 5 years
  * All-cause mortality
  * All stroke (disabling and non-disabling)
  * Hospitalization for valve-related symptoms or worsening congestive heart failure
Clinical efficacy | 30 days through 5 years
  • NYHA Class III or IV
Clinical efficacy | 30 days through 5 years
  • Prosthetic heart valve dysfunction (mean aortic valve gradient ≥20mm Hg, EOA ≤0.9-1.1cm2 [depending on body surface area] and/or DVI <0.35, AND/OR moderate or severe prosthetic valve regurgitation)
Time-related Valve Safety | 5 years
  • Structural valve deterioration:
  * Valve-related dysfunction (mean aortic valve gradient (mean aortic valve gradient ≥20mmHg, EOA ≤0.9-1.1cm2 [depending on body surface area] and/or DVI <0.35, AND/OR moderate or severe prosthetic valve regurgitation)
  * Requiring repeat procedure (TAVR or SAVR)
Time-related Valve Safety | 5 years
  * Prosthetic valve endocarditis
  * Prosthetic valve thrombosis
  * Thromboembolic events (e.g., stroke)
  * VARC bleeding, unless clearly unrelated to valve therapy (e.g., trauma)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Naber, MD, Principal Investigator — Elisabeth Krankenhaus Essen GmbH
Locations (2):
- Elisabeth Krankenhaus, Essen, Germany
- Ospedale Niguarda Ca' Granda, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: sponsor website — http://www.directflowmedical.com